CLINICAL TRIAL: NCT04104620
Title: Autoimmunity Family Background in Neurological Syndromes With Antibodies Against Glutamic-acid Decarboxylase
Brief Title: Autoimmunity in Patients With GAD-Ab and Their Relatives
Acronym: FamilyGAD
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: FamilyGAD
Record Dates: First submitted 2019-09-24; First posted 2019-09-26 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Neurological Syndromes With GAD-Ab; Organ-specific Autoimmune Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with neurological syndromes and GAD-Ab: This is a non-interventional study involving clinical data already stored in the database of the Centre de référence des syndromes neurologiques paranéoplasiques et encéphalites auto-immunes, or collected by the referral physicians the day of ordinary consultations. No biological sample is necessary to perform this study.

SUMMARY:
A group of poorly studied immune-mediated neurological syndromes are associated with antibodies against glutamic-acid decarboxylase (GAD-Ab). GAD is the rate-limiting enzyme for the synthesis of gamma aminobutyric acid (GABA) from glutamate and is expressed by inhibitory neurons of the central nervous system. Neurological syndromes with anti-GAD antibodies (GAD-Ab) are often non-paraneoplastic. They mainly include limbic encephalitis (LE), cerebellar ataxia (CA) and stiff-person syndrome (SPS). Although the pathogenic role of GAD-Ab is controversial, most patients have high serum levels and GAD-Ab are also detected in the cerebrospinal fluid (CSF) along with other inflammatory abnormalities such as oligoclonal bands. GAD-Ab may also be present in the serum of T1DM patients, as pancreatic beta cells also express GAD, but usually at much lower titers than those of neurological patients. Organ-specific autoimmune diseases, such as T1DM and autoimmune thyroid disease, are common among patients with GAD-Ab and neurological syndromes and in their relatives, suggesting a shared genetic predisposition to autoimmune disorders. This is also supported by family reports of neurological syndromes with GAD-Ab and some HLA associations described in SPS.

The aim of this study is to describe the different autoimmune organ-specific diseases present in patients with GAD-Ab and their relatives, along with to identify families with higher aggregation of autoimmune diseases and establish potential ways of inheritability.

DETAILED DESCRIPTION:
A group of poorly studied immune-mediated neurological syndromes are associated with antibodies against glutamic-acid decarboxylase (GAD-Ab). GAD is the rate-limiting enzyme for the synthesis of gamma aminobutyric acid (GABA) from glutamate and is expressed by inhibitory neurons of the central nervous system. Neurological syndromes with anti-GAD antibodies (GAD-Ab) are often non-paraneoplastic. They mainly include limbic encephalitis (LE), cerebellar ataxia (CA) and stiff-person syndrome (SPS). Although the pathogenic role of GAD-Ab is controversial, most patients have high serum levels and GAD-Ab are also detected in the cerebrospinal fluid (CSF) along with other inflammatory abnormalities such as oligoclonal bands. GAD-Ab may also be present in the serum of T1DM patients, as pancreatic beta cells also express GAD, but usually at much lower titers than those of neurological patients. Organ-specific autoimmune diseases, such as T1DM and autoimmune thyroid disease, are common among patients with GAD-Ab and neurological syndromes and in their relatives, suggesting a shared genetic predisposition to autoimmune disorders. This is also supported by family reports of neurological syndromes with GAD-Ab and some HLA associations described in SPS.

The aim of this study is to describe the different autoimmune organ-specific diseases present in patients with GAD-Ab and their relatives, along with to identify families with higher aggregation of autoimmune diseases and establish potential ways of inheritability.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a well-known neurological syndrome associated with Gad-Ab (LE, CA, SPS)
* Patient with an CSF positive for GAD-Ab;
* Patient witn an Age > 18 years old.

Exclusion Criteria:

* Patient with absence of complete clinical data.
* Patient with CSF not tested or negative for GAD-Ab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with neurological syndromes and GAD-Ab included in the database from the Centre de référence des syndromes neurologiques paranéoplasiques et encéphalites auto-immunes, Lyon
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-09-30 (Estimated); Primary Completion 2020-08-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Autoimmune organ-specific diseases in patients with GAD-Ab and their relatives | 12 Months
  To collect the different autoimmune organ-specific diseases present in patients with GAD-Ab and their relatives

SECONDARY OUTCOMES:
Inheritability in neurological syndromes with GAD-Ab | 12 Months
  To establish potential common ways of inheritability in neurological syndromes with GAD-Ab and organ-specific autoimmune diseases

CONTACTS AND LOCATIONS:
Overall Officials: Jerome HONNORAT, phd, Principal Investigator — Centre de référence des syndromes neurologiques paranéoplasiques et encéphalites auto-immunes, Lyon, France

IPD SHARING:
Plan to Share IPD: No